CLINICAL TRIAL: NCT00854711
Title: Randomized Placebo-controlled Trial of Inhaled iNO in Acute ST-segment Elevation MI Treated by Primary Angioplasty
Acronym: ENAMOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Interventional cardiologist, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-09-AH-7009-CTIL
Record Dates: First submitted 2009-02-16; First posted 2009-03-03 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: STEMI
Keywords: ST elevated Myocardical infraction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nitric oxide (Experimental): inhaled nitric oxide 80 ppm and oxygen
  Interventions: Procedure: inhaled nitric oxide
- standart of care (Placebo Comparator): no intervention
  Interventions: Procedure: inhaled nitric oxide

INTERVENTIONS:
Procedure: inhaled nitric oxide — 80 PPM
  Other Names: iNO

SUMMARY:
Reperfusion of ischemic myocardium, termed ischemia/reperfusion during the treatment of MI may result in paradoxical myocardial injury compromising myocardial salvage and left ventricular functional recovery. Nitric oxide (NO) modulates many of the processes contributing to ischemia-reperfusion injury (IR)and inhaled NO (iNO) has been shown to decease infarct size in animal models of IR. iNO has been studied in various clinical settings and has shown promise im modulating the detrimental effects of IR. Clinical toxicity potentially associated with the use of iNO was of no apparent concern in these studies. Although controlled trials of iNO therapy in humans with acute MI have not been published, anecdotal experience indicates a beneficial impact of iNO on the hemodynamic course of patients with right ventricular MI. iNO is widely used to treat neonatal hypoxemia and acute pulmonary hypertension. iNO has been studied at this dose in various clinical settings and side effects related to its use at such doses are extremely uncommon. The effect of iNO on IR injury in patients with acute ST-segment elevation MI is unknown. The investigator intend to perform a prospective, randomized, placebo-controlled, clinical trial of iNO in patients with acute MI undergoing primary percutaneous intervention to determine whether this form of therapy can decrease infarct size and improve clinical outcomes.

DETAILED DESCRIPTION:
Eligible consenting patients will be randomly assigned to either of the 2 treatment arms using a computer-generated randomization sequence. Treatment arms: 1) Intervention group, treated with inhalation of a mixture of NO 80 ppm and oxygen; or, 2) Control group, inhalation oxygen and nitrogen (placebo). In both groups, oxygen will be administered at the minimal FiO2 required to maintain arterial oxygen saturation determined by pulse oxymetry >97%. Inhalation treatment will be given throughout the angioplasty procedure via a reservoir face mask and a dedicated respiratory circuit. Nitric oxide will be delivered using an FDA-approved device marketed in Israel under license by the Ministry of Health. The device is in routine clinical use in intensive care units, neonatal care units, and catheterization laboratories. An NO-level detector will be employed in the catheterization laboratory to monitor the ambient NO exposure of the staff.

Upon arrival in the catheterization laboratory, a 40 ml blood sample will be obtained for a full chemistry panel, lipid levels, complete blood count. Creatine kinase, creatine kinase MB fraction, and troponin I will be measured at baseline and every 4 hours following the angioplasty procedure during the first 24 hours, and then every 6 hours during the second and third days, and as clinically indicated thereafter.Methemoglobin levels will be measured at baseline, every 30 minutes throughout the interventional procedure, at procedure completion, and at 4 hours post procedure.

All patients will undergo diagnostic angiography and interventional procedures as per standard clinical practice. Post procedural pharmacotherapy, sheath removal, and deployment of hemostatic devices will be left to the discretion of the attending physicians.

Following treatment in the catheterization laboratory, medical treatment throughout hospitalization and recommendations for therapy after discharge will be left to the discretion of the attending cardiologists managing patient care on the hospital wards. These cardiologists will be blinded to the patient randomization status.

ELIGIBILITY:
Inclusion Criteria:

* Subject is over 18 years old
* Subject has an acute ST segment elevation myocardial infarction defined as the presence of ST segment elevation in at least two contiguous leads or new left bundle branch block and the presence of symptoms at rest typical of myocardial ischemia for at least 30 minutes but less than 12 hours prior to admission
* Subject is eligible for primary PCI
* Subject understands the nature of the procedure and provides written informed consent prior to the catheterization procedure
* Subject is willing to comply with pre specified follow up evaluation and can be contacted by telephone
* Subject is male or a non pregnant female
* Subject is a candidate for urgent PCIintervention for reperfusion of an infarct related artery that is totally occluded and is more than 2.5mm in diameter.

Exclusion Criteria:

* Subject is currently enrolled in another investigational study of a new drug, biologic or device at the time of study screening
* Ischemic symptom onset more than 12 hours prior to presentation
* Subject with a history of a previous Q wave myocardial infarction
* A PCI procedure of any kind within 30 days prior to the procedure.
* Subject with previously known impaired left ventricular function from any reason
* Subject with STEMI that requires treatment of the left main coronary artery during the primary PCI.
* Patients who are hemodynamically unstable (Killip class 3 or 4, mechanical ventilation, life threatening ventricular arrhythmias, patients resuscitated from cardiac arrest)
* Co-morbid condition that could limit the subject's ability to participate in the trial or to comply with follow-up requirements
* Concurrent medical condition with a life expectancy of less than 12 months.
* Documented left ventricular ejection fraction less than 45% prior to the index event
* History of cerebrovascular accident or transient ischemic attack in the last 6 months
* Known severe renal failure (serum creatinine level more than2.5 mg/dl
* History of bleeding diathesis or coagulopathy or inability or unwillingness to receive blood transfusions.
* Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel and ticlopidine, cobalt, nickel, L 605 Cobalt chromium alloy, or sensitivity to contrast media, which cannot be adequately pre-medicated
* Bleeding diathesis.
* Evidence of active gastrointestinal bleeding or a history of such bleeding that is not known to have been treated and proven to have resolved
* History of hepatitis (viral, ischemic or chemically induced), clinical jaundice, history of cirrhosis
* Subject is deemed in definite need of CABG surgery during the index hospitalization
* Recent (less than 72 hours) use of sildenafil (Viagra, Revatio), verdenafil (Lefvitra), or tadalfil (Cialis)

Angiographic exclusion criteria:

* The infarct vessel is a surgical bypass graft, clinically significant left main coronary artery disease (obstruction greater than 50 percent in the left main coronary artery) in the absence of patent bypass grafts to the left anterior descending and left circumflex arteries;
* Target lesion is located in an aorto-ostial position or within 2 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX)
* target lesion(s) with severe calcification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Infarct size assessed by measurements of myocardial biomarkers (creatine kinase [CK], CK MB, troponin I) from blood samples obtained at admission and repeatedly over the next 3 days. | 3-days post randomization

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE), defined as death, myocardial infarction (MI, Q wave and non-Q wave), emergent bypass surgery, or clinically driven target lesion(s) revascularization (TLR) (repeat PCI or CABG) at 12-months. | 12-month post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Amir S Halkin, MD, Principal Investigator — TASMC
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No